CLINICAL TRIAL: NCT04014972
Title: Clinical Features, Treatment Mode and Health Outcomes of Chest Pain Patients in China: China Chest Pain Center Accreditation Programme,CHANGE-chest Pain Research
Brief Title: Clinical Features, Treatment Mode and Health Outcomes of Chest Pain Patients in China (CHANGE)
Acronym: CHANGE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China Cardiovascular Association (Other)
Collaborators: Peking University First Hospital (Other); Shanghai Zhongshan Hospital (Other); Peking University (Other)
Responsible Party: Sponsor
Other Study IDs: GUSU19005
Record Dates: First submitted 2019-07-03; First posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Chest Pain Center; STEMI - ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Myocardial Infarction

SUMMARY:
Chinese Cardiovascular Association is an association dedicated to establishing Chest Pain Centers in hospitals that have basic qualifications and meet pre-designed quality control targets.The vision of Chinese Cardiovascular Association is the cardiovascular health of every Chinese, and the mission is to realize the early arrival of the inflection point of cardiovascular events in China.The institute of China Heart House is responsible for the daily management and implementation of Chinese Cardiovascular Association and the implementation and management of the Chest Pain Center construction project.In order to improve standard treatment and chest pain system management to achieve better outcomes for patients, China Heart House established the chest pain center database.The database includes patients in 4129 registered hospitals in 31 provinces in China who have been admitted with chest pain.The database can reflect the clinical characteristics, treatment and outcome of patients with chest pain in China.

This non-interventional, retrospective study analyzed the chest pain center database to understand the demographics, clinical characteristics, treatment patterns and clinical outcomes of patients with chest pain, and to analyze the effects of different treatment patterns, including chest pain centers and related collaborative treatment networks.The results of the study will assess the gap between the real-world situation and the recommendations of the guidelines and reflect the effect of chest pain centers and related collaborative treatment networks on the treatment process and service quality.The research results can be directly translated into the basis of medical treatment system intervention, and also provide decision-making reference for improving the certification standards and quality control of chest pain centers.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and above
* patients admitted with chest pain
* diagnosis is made by the treating physician based on local practice and clinical judgment

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was inpatients (18 years and older) admitted to the Chest Pain Central database with symptoms of chest pain.The database registration of this study was conducted in 4129 registered hospitals in 31 provinces in China.All hospitals participating in the Chest Pain Center program are encouraged to manage patients in accordance with local standard practices (as recommended by current Chinese guidelines).
  This study will include data on all patients in the chest pain central database.
Sampling Method: Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
mean and standard deviation of STEMI (ST-segment elevated Myocardial Infarction)patients | baseline
  mean and standard deviation of STEMI patients
Proportion of STEMI (ST-segment elevated Myocardial Infarction)patients | baseline
  Proportion of female STEMI patients
emergency information of STEMI patients | baseline
  Path to hospital
  First medical contact time
  Does the patient circumvent emergency
  Telecardiogram transmission
  STEMI Reperfusion Therapy
  Initiation time of interventional surgery
  Catheter chamber activation time
  Time of arrival of patient in catheter room
  Guide wire passage time
  D2B time
admission status of STEMI patients | baseline
  admission status of STEMI patients
hospitalization evaluation of STEMI patients | baseline
  value of serum troponin and serum creatinin of STEMI patients
In-hospital mortality of STEMI patients | baseline
  In-hospital mortality of STEMI patients
Hospitalization days of STEMI patients | baseline
  Hospitalization days of STEMI patients
Total cost of STEMI patients | baseline
  Total cost of STEMI patients